CLINICAL TRIAL: NCT02837328
Title: Magnesium Supplementation for the Prevention of Supraventricular Arrhythmias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1605M87323
Record Dates: First submitted 2016-06-22; First posted 2016-07-19 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Premature Atrial Contraction
Keywords: Magnesium Supplementation; Magnesium; Dietary Supplement; Arrhythmia
MeSH Terms: conditions — Atrial Premature Complexes; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Magnesium Supplement (Experimental): 400 mg Magnesium Citrate 1x daily for 12 weeks
  Interventions: Drug: Oral Magnesium Supplement
- Placebo (Placebo Comparator): Placebo pill resembling 400 mg Magnesium Citrate 1x daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Magnesium Supplement — 400 mg Magnesium Citrate 1x daily for 12 weeks
  Arms: Oral Magnesium Supplement
Drug: Placebo — Placebo pill resembling 400 mg Magnesium Citrate 1x daily for 12 weeks
  Arms: Placebo

SUMMARY:
The primary objective of this research is to determine whether oral magnesium supplementation in healthy, community-living individuals will be associated with reductions in the burden of arrhythmias in the upper chambers of the heart (supraventricular arrhythmias).

DETAILED DESCRIPTION:
To evaluate the primary objective, the Investigator will conduct a double-blind randomized trial assigning participants to receive 400 mg of oral magnesium in the form of magnesium citrate once daily or placebo. The investigators will recruit 60 individuals 55 years of age and older without a prior history of cardiovascular disease. At baseline, participants will undergo a basic examination, answer questionnaires and provide a blood sample to determine circulating magnesium levels. Participants will then wear an FDA-approved heart rhythm monitor (Zio ® XT Patch) for 2 weeks. At the end of 2 weeks they will begin taking their assigned treatment (magnesium or placebo), and will continue doing so for a total of 12 weeks (through study week 14). After 10 weeks of taking the supplement or placebo (study week 12), they will have a final study visit in which the participants will provide another blood sample for assessment of circulating magnesium, and will be asked to wear the heart rhythm monitor for another 2 weeks (through study week 14). The primary endpoint will be the change in burden of premature atrial contractions (PACs), measured in episodes per day, between baseline and final follow-up visit. A secondary outcome will be the change in circulating magnesium between both exams.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 and older
* Ability to speak English
* Availability to attend baseline and follow-up visit approximately 12 weeks after baseline

Exclusion Criteria:

* Prior history of heart disease (coronary heart disease, heart failure, atrial fibrillation), stroke, severe renal disease
* Use of type I and III antiarrhythmics or digoxin
* Current use of magnesium supplements
* Any prior history of allergy or intolerance to magnesium
* Prior history of inflammatory bowel disease or any severe gastrointestinal disorder

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Lutsey, PhD, Principal Investigator — University of Minnesota; Alvaro Alonso, MD PhD, Principal Investigator — University of Minnesota; Lin Y Chen, MD, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota - Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alonso A, Chen LY, Rudser KD, Norby FL, Rooney MR, Lutsey PL. Effect of Magnesium Supplementation on Circulating Biomarkers of Cardiovascular Disease. Nutrients. 2020 Jun 6;12(6):1697. doi: 10.3390/nu12061697. PMID 32517192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants of 55 years of age or older were recruited using fliers, the University of Minnesota StudyFinder website, invitations to individuals enrolled in the ResearchMatch research volunteer database, and invitations to University of Minnesota School of Public Health employees.
Pre-assignment Details: Participants attended a baseline visit where measurements were conducted and a Zio XT Patch heart rhythm monitor was applied by trained staff. After wearing the patch for 2 weeks, the participants were randomized 1:1 to either magnesium oxide or a placebo using block randomization within two strata of age (younger than 65 and 65 and older).
Period: Overall Study
Arm/Group | Oral Magnesium Supplement | Placebo
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Magnesium Supplement | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (5.3) | 61.6 (5.2) | 61.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 4 | 12 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 27 | 29 | 56
  Race/Ethnicity: Non-White | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59
Serum Magnesium Concentrations [Mean (Standard Deviation); unit: mEq/L] | 1.74 (0.12) | 1.71 (.1) | 1.72 (0.11)
Premature Arterial Contractions Burden [Mean (Standard Deviation); unit: episode/hour] | 8.5 (14) | 20.2 (80) | 14.5 (58)
Log Premature Arterial Contractions Burden [Mean (Standard Deviation); unit: log(Episodes/hour)] | 1.26 (1.35) | 1.04 (1.49) | 1.15 (1.42)

OUTCOME MEASURES:

1. Primary Outcome: Change in Premature Atrial Contractions (PACs)
Description: The primary endpoint will be the change in burden of PACs
Time Frame: Change from Baseline at 10 weeks
Measure: Mean (Standard Deviation); unit: Episodes/hour
Arm/Group | Oral Magnesium Supplement | Placebo
Number analyzed (Participants) | 29 | 30
Episodes/hour | -0.6 (7) | -5.6 (33)

2. Secondary Outcome: Change in Magnesium Concentration
Description: The secondary endpoint will be the change in circulating magnesium between baseline and a follow-up visit 10 weeks later.
Time Frame: Baseline and week 10
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Oral Magnesium Supplement | Placebo
Number analyzed (Participants) | 29 | 30
mEq/L | 0.07 (0.09) | 0 (.1)

ADVERSE EVENTS:
Time Frame: 59 days, from day 21 of the intervention to day 80
Description: Participants were asked an open-ended question about the occurrence of adverse events. Adverse event information was collected in such a way that individual adverse event terms cannot be separated.
Arm/Group | Oral Magnesium Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 15/29 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Magnesium Supplement (N=29) | Placebo (N=30)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 15 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT02837328/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT02837328/SAP_001.pdf